CLINICAL TRIAL: NCT07218861
Title: You Belong and You Matter: An Exploration of Self-injurious Thoughts and Behaviors in LGTBQ+ Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ULouisville
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Supportive Messages; Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive Message Condition (Experimental): Supportive messages
  Interventions: Behavioral: Supportive Messages
- No Message Control (No Intervention): Control

INTERVENTIONS:
Behavioral: Supportive Messages — Participants received 28 supportive messages (2 per day) for 14 days
  Arms: Supportive Message Condition

SUMMARY:
Individuals with minoritized sexual and gender identities (i.e., LGBTQ+ individuals) are at a greater risk for self-injurious thoughts and behaviors than their cisgender, straight peers (Haas et al., 2010; Liu et al., 2017; Gorse, 2022). There is a dearth of empirically supported interventions for self-injurious thoughts and behaviors (Linehan, 2008; Riblet et al., 2017), and those that exist are not tailored to people in the LGBTQ+ community (Gorse, 2022; Haas et al., 2010). Therefore, the aim of this study is to test the effectiveness of a brief LGBTQ+ affirming text message intervention in reducing self-injurious thoughts and behaviors among LGBTQ+ individuals.

DETAILED DESCRIPTION:
Scope of the work

LGBTQ+ individuals are at a greater risk for self-injurious thoughts and behaviors than their cisgender, straight peers. Despite this known risk, there are no culturally sensitive empirically supported treatments for self-injurious thoughts and behaviors for LBGTQ+ individuals. Therefore, the aim of this study is to test the effectiveness of a brief LGBTQ+ affirming text message intervention in reducing self-injurious thoughts and behaviors among LGBTQ+ individuals. Participants will be 100 LGBTQ+ adults who report self-injurious thoughts and/or behaviors in the last month. All participants will do 14 days of ecological momentary assessment (brief assessments on their mobile device 5 times a day) pre-randomization. After this period, half the participants will receive 2 brief affirming messages a day (morning and afternoon) for 14 days, and half of the participants will receive no messages for 14 days. The text messages will be designed to communicate belonging and importance for LGBTQ+ individuals in society (e.g., "There are over 9,000,000 LGBTQ+ people in the United States. You are not alone". Then all participants will complete another 14 days of ecological momentary assessment. During the assessment periods, participants will report on experiences of discrimination, belongingness, perceived burdensome, and self-injurious thoughts. We predict that participants in the mobile health condition will have a significant decrease in self-injurious thoughts and behaviors from pre- to post-intervention, whereas there will be no change in the control condition. We also predict that participants in the mobile health condition will lead to a significant decrease in thwarted belongingness and perceived burdensomeness. Finally, we predict that our intervention will help break the link between of experiences discrimination and self-injurious thoughts and behaviors by reducing feelings of thwarted belongingness and perceived burdensomeness in response to sexual and gender minority stress. If the effectiveness of our intervention is supported by the data, this intervention could be scaled up and be made available to the LGBTQ+ community broadly.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years or older b) have an LGBTQ+ identity (e.g., a sexual orientation other than exclusively straight and/or a gender identity other than exclusively cisgender) c) report at least one self-injurious thought (e.g., suicidal or nonsuicidal self-injury ideation), or behavior (nonsuicidal self-injury, suicide attempt) in the last month

Exclusion Criteria:

* Younger than 18, exclusivilty cisgender, heterosexual, no history of SITB in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Self-injurious thoughts and behavior | last two hours
  self reported

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided